CLINICAL TRIAL: NCT01127438
Title: A Double-blind, Randomized, Multicenter, Dose-ranging Study to Evaluate the Safety and Efficacy of LUSEDRA (Fospropofol Disodium) as an Intravenous Sedative for Diagnostic or Therapeutic Colonoscopy in Adult Special Populations
Brief Title: A Dose-ranging Study to Evaluate the Safety and Efficacy of LUSEDRA (Fospropofol Disodium) as an Intravenous Sedative for Diagnostic or Therapeutic Colonoscopy in Adult Special Populations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2083-A001-406
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Sedation
Keywords: Monitored anesthesia care sedation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- fospropofol disodium Subgroup 1 Lower Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 1 Lower Dose
- : fospropofol disodium Subgroup 1 Approved Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 1 Approved Dose
- fospropofol disodium Subgroup 2 Lower Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 2 Lower Dose
- fospropofol disodium Subgroup 2 Approved Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 2 Approved Dose
- fospropofol disodium Subgroup 3 Lower Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 3 Lower Dose
- fospropofol disodium Subgroup 3 Approved Dose (Active Comparator)
  Interventions: Drug: fospropofol disodium Subgroup 3 Approved Dose

INTERVENTIONS:
Drug: fospropofol disodium Subgroup 1 Lower Dose — Dose of Initial IV (Titration) Bolus 6.5mg/kg) (administered to Subgroup 1, Weight < 60 kg and Age < 65 years and ASAI and II)
  Arms: fospropofol disodium Subgroup 1 Lower Dose
Drug: fospropofol disodium Subgroup 1 Approved Dose — (Dose of Initial IV (Titration) Bolus 385mg) (Administered to Subgroup 1, Weight <60 kg and Age <65 years and ASAI and II)
  Arms: : fospropofol disodium Subgroup 1 Approved Dose
Drug: fospropofol disodium Subgroup 2 Lower Dose — Dose of Initial IV (Titration) Bolus 4.875 mg/kg) (administered to Subgroup 2, Weight < 60 kg and Age >/=65 years and ASA 3 or 4
  Arms: fospropofol disodium Subgroup 2 Lower Dose
Drug: fospropofol disodium Subgroup 2 Approved Dose — (Dose of Initial IV (Titration) Bolus 297.5mg) (Administered to Subgroup 2, Weight <60 kg and Age >/=65 years and ASA 3 or 4
  Arms: fospropofol disodium Subgroup 2 Approved Dose
Drug: fospropofol disodium Subgroup 3 Lower Dose — (Dose of Initial IV (Titration) Bolus 3.9mg/kg) (Administered to Subgroup 3, Weight >/= 60 kg and Age >/= 65 years and ASA 3 or 4
  Arms: fospropofol disodium Subgroup 3 Lower Dose
Drug: fospropofol disodium Subgroup 3 Approved Dose — Dose of Initial IV (Titration) Bolus 4.875 mg/kg) (Administered to Subgroup 3, Weight >/= 60 kg and Age >/= 65 years and ASA 3 or 4
  Arms: fospropofol disodium Subgroup 3 Approved Dose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of LUSEDRA (fospropofol disodium) and to determine whether a dose lower than currently approved can provide effective moderate sedation required to complete diagnostic or therapeutic procedures.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, parallel-group, multicenter, dose-ranging study, in age >/= 65 years, and/or weight < 60 kg, and/or American Society of Anesthesiologists (ASA) Physical Classification Status 3 or 4 subjects using either the approved dose modification or 1 lower dose, to achieve a moderate level of sedation required to complete the scheduled diagnostic or therapeutic procedure. Three subgroups of subjects will be included. For Subgroup 1 and Subgroup 2, approximately equal numbers of subjects will be enrolled into 2 strata: weight >/= 55 kg and weight < 55 kg. For Subgroup 1 and Subgroup 2, subjects will be randomly assigned to 1 of 2 dose groups in a 1:1 ratio within each stratum. For Subgroup 3, subjects will be randomly assigned to 1 of 2 dose groups in a 1:1 ratio.

ELIGIBILITY:
Subjects who meet all of the following criteria will be included in the study:

1. Male and female adult candidates for diagnostic or therapeutic colonoscopy with at least one of the following characteristics:

   * Subgroup 1: Weight < 60 kg and age >/= 18 to < 65 years and ASA I or II;
   * Subgroup 2: Weight < 60 kg and age >/= 65 years and/or ASA 3 or 4; or
   * Subgroup 3: Weight >/=60 kg and age >/= 65 years and/or ASA 3 or 4.
2. Females of childbearing potential must have a negative beta human chorionic gonadotropin (?hCG) urine pregnancy test at Visit 1 (Screening) and prior to starting study drug (Visit 2). Female subjects of childbearing potential must agree to be abstinent or to use a highly effective methods of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine device [IUD], or have a vasectomised partner) having starting for at least 1 menstrual cycle prior to starting study drug and throughout the entire study period and for 30 days after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential;
3. Are willing and able to comply with all aspects of the protocol; and
4. Provide written informed consent.

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Females who are pregnant (positive BhCG urine pregnancy test) or breastfeeding;
2. Subjects who do not meet nil per os (NPO) requirement of no solid foods within 8 hours and clear fluids up to 3 hours before the procedure (assessed only at Baseline);
3. Evidence of clinically significant disease or a history of a concomitant medical condition (eg, cardiac, respiratory, gastrointestinal, renal disease) that, in the opinion of the Investigator, could affect the subject's safety or ability to safely complete the study;
4. Subjects with hypersensitivity to LUSEDRA or any other components of LUSEDRA, including its active metabolite, propofol;
5. History of drug or alcohol dependency or abuse within approximately the last 2 years; or
6. The Investigator believes to be medically unfit to receive the study drug or unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Ferry, Study Director — Eisai Inc.
Locations (23):
- United States (23):
  - Hope Research Institute, Phoenix, Arizona
  - Southern California Permanente Medical Group, Baldwin Park, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Center for Advanced Gastroenterology, Maitland, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Sheridan Clinical Research, Sunrise, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Creighton University Medical Center, Omaha, Nebraska
  - Research Associates of New York, LLP, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University Medical Center Department of Anesthesiology, Columbus, Ohio
  - Ilumina Clinical Associates, Keystone Headache and Pain Mgt Center, Tyrone Hospital, Tyrone, Pennsylvania
  - Ilumina Clinical Associates, Uniontown, Pennsylvania
  - Digestive Health Associates, Plano, Texas
  - Clinical Trial Network, Spring, Texas
  - Utah Digestive Health Institute, Clinton, Utah
  - Northern Utah Gastroenterology, Logan, Utah
  - Advance Clinical Research, Odgen, Utah
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Subgroup 1, Lower Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 18 years but below 65 years, and an American Society of Anesthesiologists (ASA) physical classification status 1 or 2. The doses were weight-adjusted for each subject, with 6.5mg of Lusedra per kg during the Randomization Phase (1 day).
- Subgroup 1, Approved Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 18 years but below 65 years, and an American Society of Anesthesiologists (ASA) physical classification status 1 or 2. A dose of 385mg of Lusedra was taken during the Randomization Phase (1 day).
- Subgroup 2, Lower Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiologists (ASA) physical classification status 3 or 4. The doses were weight-adjusted for each subject, with 4.875mg of Lusedra per kg during the Randomization Phase (1 day).
- Subgroup 2, Approved Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiologists (ASA) physical classification status 3 or 4. A dose of 297.5mg of Lusedra was taken during the Randomization Phase (1 day).
- Subgroup 3, Lower Dose: This arm consisted of subjects with a weight at or above 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiologists (ASA) physical classification status 3 or 4. The doses were weight-adjusted for each subject, with 3.9mg of Lusedra per kg during the Randomization Phase (1 day).
- Subgroup 3, Approved Dose: This arm consisted of subjects with a weight at or above 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiologists (ASA) physical classification status 3 or 4. The doses were weight adjusted for each subject, with 4.875mg of Lusedra per kg during the Randomization Phase (1 day).
Period: Overall Study
Arm/Group | Subgroup 1, Lower Dose | Subgroup 1, Approved Dose | Subgroup 2, Lower Dose | Subgroup 2, Approved Dose | Subgroup 3, Lower Dose | Subgroup 3, Approved Dose
Started | 25 | 25 | 26 | 24 | 28 | 25
Completed | 25 | 25 | 26 ((n=25) One subject randomized to the approved dose group received a lower dose in error.) | 24 ((n=25) One subject randomized to the approved dose group received a lower dose in error.) | 28 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subgroup 1, Lower Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 18 years but below 65 years, and an American Society of Anesthesiolog ists (ASA) physical classification status 1 or 2. The doses were weightadjusted for each subject, with 6.5mg of Lusedra per kg during the Randomizatio n Phase (1 day).
- Subgroup 1, Approved Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 18 years but below 65 years, and an American Society of Anesthesiolog ists (ASA) physical classification status 1 or 2. A dose of 385mg of Lusedra was taken during the Randomizatio n Phase (1 day).
- Subgroup 2, Lower Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiolog ists (ASA) physical classification status 3 or 4. The doses were weightadjusted for each subject, with 4.875mg of Lusedra per kg during the Randomizatio n Phase (1 day).
- Subgroup 2, Approved Dose: This arm consisted of subjects with a weight below 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiolog ists (ASA) physical classification status 3 or 4. A dose of 297.5mg of Lusedra was taken during the Randomizatio n Phase (1 day).
- Subgroup 3, Lower Dose: This arm consisted of subjects with a weight at or above 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiolog ists (ASA) physical classification status 3 or 4. The doses were weightadjusted for each subject, with 3.9mg of Lusedra per kg during the Randomizatio n Phase (1 day).
- Subgroup 3, Approved Dose: This arm consisted of subjects with a weight at or above 60kg, an age at or greater than 65 years, and/or an American Society of Anesthesiolog ists (ASA) physical classification status 3 or 4. The doses were weightadjusted for each subject, with 4.875mg of Lusedra per kg during the Randomizatio n Phase (1 day).
- Total: Total of all reporting groups
Arm/Group | Subgroup 1, Lower Dose | Subgroup 1, Approved Dose | Subgroup 2, Lower Dose | Subgroup 2, Approved Dose | Subgroup 3, Lower Dose | Subgroup 3, Approved Dose | Total
Number analyzed (Participants) | 25 | 25 | 26 | 24 | 28 | 25 | 153
Age, Customized [Number; unit: Participants] — Safety Analysis Set.
  Participants
    <65 Years | 25 | 25 | 6 | 8 | 8 | 5 | 77
    >=65 Years | 0 | 0 | 20 | 16 | 20 | 20 | 76
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Analysis Set: All subjects who received atleast one dose of study medication and had atleast one postdose safety assessment.
  Participants
    Female | 25 | 24 | 23 | 21 | 13 | 9 | 115
    Male | 0 | 1 | 3 | 3 | 15 | 16 | 38
Race/Ethnicity, Customized [Number; unit: Participants] — Safety Analysis Set.
  Participants
    White | 20 | 21 | 19 | 20 | 22 | 25 | 127
    Black or African American | 1 | 2 | 2 | 1 | 5 | 0 | 11
    Asian | 3 | 2 | 4 | 3 | 1 | 0 | 13
    American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Other | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sedation Success
Description: Sedation success was defined as subjects who met the following 4 criteria: had 3 consecutive Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores at or less than 4 after administration of sedative medication, completed the procedure, did not require the use of alternative sedative medication, and did not require manual/mechanical ventilation. The MOAA/S score was used to clinically rate the level of sedation using a score of 0 to 5 based on the subject's level of responsiveness. A high score on the MOAA/S scale indicated a lower level of sedation.
Time Frame: Day 1
Population: Full Analysis Population: All treated subjects who received study drug and had at least one postdose efficacy measurement.
Measure: Number; unit: Participants
Arm/Group | Subgroup 1, Lower Dose | Subgroup 1, Approved Dose | Subgroup 2, Lower Dose | Subgroup 2, Approved Dose | Subgroup 3, Lower Dose | Subgroup 3, Approved Dose
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 28 | 25
Participants | 18 | 24 | 18 | 21 | 19 | 24

2. Secondary Outcome: Number of Participants With Treatment Success
Description: Treatment success was defined as subjects who met the following 3 criteria: completed the procedure, did not require the use of alternative sedative medication, and did not require manual/mechanical ventilation.
Time Frame: Day 1
Population: Full Analysis Population.
Measure: Number; unit: Participants
Arm/Group | Subgroup 1, Lower Dose | Subgroup 1, Approved Dose | Subgroup 2, Lower Dose | Subgroup 2, Approved Dose | Subgroup 3, Lower Dose | Subgroup 3, Approved Dose
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 28 | 25
Participants | 18 | 24 | 18 | 21 | 19 | 24

3. Secondary Outcome: Number of Participants With Modified Sedation Success
Description: Modified sedation success was defined as a subject who was a sedation success and did not have a MOAA/S score <2 any time after administration of sedative medication. Sedation success was defined as subjects who had 3 consecutive MOAA/S scores at or less than 4 after administration of sedative medication, completed the procedure, did not require the use of alternative sedative medication, and did not require manual/mechanical ventilation. The MOAA/S score was used to clinically rate the level of sedation using a score of 0 to 5 based on the level of responsiveness.
Time Frame: Day 1
Population: Full Analysis Population.
Measure: Number; unit: Participants
Arm/Group | Subgroup 1, Lower Dose | Subgroup 1, Approved Dose | Subgroup 2, Lower Dose | Subgroup 2, Approved Dose | Subgroup 3, Lower Dose | Subgroup 3, Approved Dose
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 28 | 25
Participants | 16 | 20 | 18 | 18 | 17 | 20

ADVERSE EVENTS:
Description: The AE/SAE information reflects the Safety Population for the intended randomization and does not redistribute the one subject randomized to the lower dose group in error.
Groups:
- Lower Dose; Approved Dose: Includes subgroups 1-3
Arm/Group | Lower Dose | Approved Dose
Serious Adverse Events (participants affected / at risk) | 1/79 | 2/74
Other Adverse Events (participants affected / at risk) | 23/79 | 15/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lower Dose (N=79) | Approved Dose (N=74)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lower Dose (N=79) | Approved Dose (N=74)
Diverticulum (Gastrointestinal disorders) | 8 | 2
Polyp (General disorders) | 5 | 2
Burning Sensation (Nervous system disorders) | 6 | 2
Paraesthesia (Nervous system disorders) | 5 | 4
Pruritus Genital (Reproductive system and breast disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No